CLINICAL TRIAL: NCT07029035
Title: Evaluation of the Clinical and Biochemical Efficacy of Repeated Injectable Platelet-Rich Fibrin Application Following Scaling and Root Planing in Patients With Periodontitis
Brief Title: Evaluation of Repeated Injectable PRF Following SRP in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Health Sciences University-Scientific Research Projects Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/254
Record Dates: First submitted 2025-05-28; First posted 2025-06-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis Stage III
Keywords: Tgf-β; Prf; Pf 4; Periodontitis; Pdgf; Split mouth; Mpo; İ-prf
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: This study utilized a split-mouth, within-subject design rather than a classical crossover or parallel group design. Each subject received both the intervention (PRF) and control (no PRF) on different sites of the oral cavity.
Who Masked: Participant
Masking Description: In addition to masking the participants, the researcher who performed the biochemical analyses was also masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Site (Experimental): Repeated application of İ-PRF to periodontal pockets in the test sites.
  Interventions: Biological: İnjectable platelet-rich fibrin
- Control Site (Sham Comparator): Control sites received a sham intervention consisting of sterile saline solution irrigation into the periodontal pockets, to mimic the procedural aspects of PRF placement without delivering any biologically active material.
  Interventions: Other: Sterile saline (0.9%)

INTERVENTIONS:
Biological: İnjectable platelet-rich fibrin — Repeated application of I-PRF to the periodontal pockets in the test sites was performed twice: once immediately following scaling and root planing (SRP), and once at the third week.
  Arms: Test Site
Other: Sterile saline (0.9%) — Control sites received a sham intervention consisting of sterile saline solution irrigation into the periodontal pockets, to mimic the procedural aspects of PRF placement without delivering any biologically active material.
  Arms: Control Site

SUMMARY:
The goal of this clinical trial is to learn if a treatment called injectable platelet-rich fibrin (i-PRF) helps improve gum health in people with a type of gum disease called Stage 3 Grade B periodontitis.

The main questions this study aims to answer are:

Does i-PRF help reduce gum inflammation and support healing? Are there changes in certain biological markers after using i-PRF? Researchers will compare two sides of the mouth. One side will receive i-PRF, and the other will be treated with salt water (saline) as a comparison.

Participants will:

Have a dental cleaning called scaling and root planing (SRP) Get i-PRF injected into deep gum pockets on one side of the mouth Have salt water placed in the other side's gum pockets Give gum fluid samples and have gum measurements taken at several visits (including 3 months later) Provide a small blood sample to prepare the i-PRF Researchers will collect and study gum fluid and look at markers related to healing and inflammation. The study will help find out if i-PRF is useful as a new treatment option for gum disease.

DETAILED DESCRIPTION:
A total of 20 patients diagnosed with Stage 3 Grade B Periodontitis based on clinical and radiographic findings will be included in this study at the Department of Periodontology, Faculty of Dentistry, Gülhane University. Eligible participants will be systemically healthy, non-smokers, not pregnant or breastfeeding, not on any medications, and must not have received any periodontal treatment or antibiotics within the past six months.

All participants will be informed about the study in detail, and written and verbal informed consent will be obtained from those who voluntarily agree to participate.

The study will be designed as a randomized controlled split-mouth clinical trial, in which the periodontal pockets in one half of the mouth will serve as the test site, and those in the other half will serve as the control site. Allocation of test and control sides will be determined by coin toss. Baseline and 3-month clinical periodontal parameters - including Plaque Index (PI), Gingival Index (GI), Bleeding on Probing (BOP), Probing Pocket Depth (PPD) and Clinical Attachment Level (CAL) will be recorded using a Williams periodontal probe.

For biochemical analysis, gingival crevicular fluid (GCF) samples will be collected from the deepest periodontal pockets at the test and control sites at four time points: baseline, 7 days after the first application of injectable platelet-rich fibrin (i-PRF), 7 days after the second application, and at 3 months. GCF collection will be performed using Periopaper strips after isolating the area with cotton rolls and gently removing supragingival plaque. Strips will be inserted into the pocket until resistance is felt, held in place for 15 seconds, and then analyzed for volume using a Periotron device. Samples will then be stored in Eppendorf tubes at -80°C until biochemical analysis. Levels of Platelet Factor-4 (PF-4), Myeloperoxidase (MPO), Transforming Growth Factor Beta (TGF-β), and Platelet-Derived Growth Factor (PDGF) in GCF will be analyzed using ELISA.

Following baseline measurements and GCF sampling, scaling and root planing (SRP) will be performed in two sessions, spaced one week apart, using standard ultrasonic and hand instruments (curettes and Gracey curettes).Venous blood samples (15 ml) will be drawn from the antecubital vein using sterile syringes and transferred into two plain tubes. The samples will be centrifuged at 1000 rpm for 3 minutes. The injectable platelet-rich fibrin (i-PRF) from the upper layer will be collected using a 5 ml syringe and administered into all deep periodontal pockets (≥4 mm) in the test quadrant. The application will be followed by gentle digital compression with a gauze sponge for 1 minute to allow polymerization and retention of the material.

In the control quadrant, deep pockets will be irrigated with sterile saline solution and similar digital compression will be applied to ensure blinding of the participants to the allocation. On the third week, the procedure will be repeated: i-PRF will be reapplied to the test sites, and saline irrigation will be repeated for the control sites. At the 3-month follow-up, all clinical indices will be reassessed, and last GCF samples will be collected.

Statistical Analysis:

All data will be analyzed using SPSS for Windows, Version 26.0 (SPSS Inc., USA). Descriptive statistics will be presented as mean ± standard deviation for continuous variables. The Shapiro-Wilk test will be used to assess the normality of data distribution. Differences between test and control sites and between time points will be analyzed using the paired samples t-test or Wilcoxon signed-rank test, depending on data distribution. A p-value of <0.05 will be considered statistically significant.

A power analysis, based on a similar previous study, indicated that including 20 test and 20 control samples (a total of 40 sites) would provide 98% statistical power.

An application will be submitted to the Scientific Research Projects Coordination Unit (BAP) to support the study with required materials and kits.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Stage 3 Grade B periodontitis
* Being between the ages of 18-65

Exclusion Criteria:

* Smoking
* Having a systemic disease
* Taking any medication
* Being pregnant or breastfeeding
* Having received chemotherapy, radiotherapy or immunosuppressant treatments
* Having received periodontal treatment in the last 6 months
* Having used antibiotics in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in GCF levels of TGF-β and PDGF at multiple time points. | From baseline to third month
  Biochemical markers will be analyzed at baseline, 2 weeks, 4 weeks, and 3 months. The biochemical data will be correlated with clinical periodontal parameters to assess the relationship between molecular changes and clinical outcomes, thereby providing a comprehensive evaluation of treatment efficacy.
Changes in clinical periodontal parameters, including Probing Pocket Depth and Clinical Attachment Level, will be evaluated at baseline and at the third month. | From baseline to third month
  Clinical data will be evaluated at baseline and at the third month.

SECONDARY OUTCOMES:
Changes in GCF levels of PF 4 and MPO at multiple time points. | From baseline to third month
  Clinical data will be evaluated at baseline and at the third month, while biochemical markers will be analyzed at baseline, 2 weeks, 4 weeks, and 3 months. The biochemical data will be correlated with clinical periodontal parameters to assess the relationship between molecular changes and clinical outcomes, thereby providing a comprehensive evaluation of treatment efficacy.
Changes in clinical periodontal parameters, including Plaque Index, Gingival Index, and Bleeding on Probing evaluated at baseline and at the third month. | From baseline to third month
  Clinical data will be evaluated at baseline and at the third month.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi Gulhane Dis Hekimligi Fakultesi, Ankara, Turkey (Türkiye)